CLINICAL TRIAL: NCT05715632
Title: Prospective, Single Arm, Single Center Exploratory Study on the New Adjuvant Therapy of Camrelizumab Combined With XELOX Regimen for Locally Advanced Gastric Cancer
Brief Title: New Adjuvant Treatment of Locally Advanced Resectable Gastric Cancer With Carelizumab and XELOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202108-20
Record Dates: First submitted 2022-12-21; First posted 2023-02-08 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carrelizumab combined with XELOX (Experimental): Before surgery, the patient received standard dose of Carrelizumab combined with XELOX regimen for 4 courses of treatment, and within 3-4 weeks after the completion of the fourth administration, preoperative imaging examination was conducted to evaluate the efficacy of new adjuvant treatment and the possibility of radical D2 resection, and to receive radical surgery for gastric cancer
  Interventions: Drug: Carrelizumab combined with XELOX

INTERVENTIONS:
Drug: Carrelizumab combined with XELOX — Before surgery, the patient received standard dose of carrelizumab combined with XELOX regimen for 4 courses of treatment, and within 3-4 weeks after the completion of the fourth administration, preoperative imaging examination was conducted to evaluate the efficacy of new adjuvant treatment and the possibility of radical D2 resection, and to receive radical hand surgery for gastric cancer

SUMMARY:
To evaluate the efficacy and safety of carelizumab combined with XELOX regimen in neoadjuvant treatment of locally advanced resectable gastric cancer

DETAILED DESCRIPTION:
This study is a prospective, single center, single arm clinical study. This study plans to include 67 patients with locally advanced gastric adenocarcinoma who can be operated without any treatment as the study object. After signing the informed consent, they are screened to meet the inclusion criteria. After receiving the standard dose of karelizumab combined with XELOX regimen for 4 courses of treatment before surgery, and within 3-4 weeks after the completion of the fourth administration, preoperative imaging examination is used to evaluate the efficacy of new adjuvant treatment and the possibility of radical D2 resection, The patient received radical surgical treatment for gastric cancer, and continued to receive adjuvant treatment of the original scheme after the operation (the first treatment started 6 weeks ± 2 weeks after the operation, and can not exceed 3 months).

ELIGIBILITY:
Inclusion Criteria:

* Sign the written informed consent before implementing any test related process
* Endoscopic or enhanced CT /MRI scanning (combined with ultrasonic gastroscopy and diagnostic laparoscopic exploration if necessary) cTNM was diagnosed as cT3-4aN1-3M0, and the investigator assessed that the lesion was resectable;
* Have not received systematic treatment for current diseases in the past, including surgical treatment, anti-tumor radiotherapy and chemotherapy /immunotherapy;
* Patients who agree to receive radical surgical treatment and have no surgical contraindication as judged by the surgeon
* ECOG score 0-1;
* The expected survival time is more than 6 months;
* Female subjects of childbearing age should receive urine or serum pregnancy test within 3 days before receiving the first study drug (the first day of the first cycle) and the result is negative. If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Women of non childbearing age are defined as those who have had at least one year after menopause, or who have undergone surgical sterilization or hysterectomy;
* If there is a risk of pregnancy, all subjects (male or female) should use contraceptives with an annual failure rate of less than 1% during the whole treatment period until 120 days after the last study drug administration (or 180 days after the last chemotherapy drug administration)

Exclusion Criteria:

* Other malignant diseases (excluding skin basal cell carcinoma, skin squamous cell carcinoma, and /or carcinoma in situ after radical resection) diagnosed within 5 years before the first administration;
* Known endoscopic signs of active hemorrhage of the lesion;
* Currently participating in the intervention clinical research treatment, or receiving other research drugs or using research instruments within 4 weeks before the first administration;
* Have received the following therapies in the past: anti PD-1, anti PD-L1 or anti PD-L2 drugs or drugs targeting another kind of stimulation or synergistic inhibition of T cell receptor (including but not limited to CTLA-4, OX-40, CD137, etc.);
* Within 2 weeks before the first administration, he has received systematic systemic treatment with Chinese patent medicine with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except for local use to control pleural effusion);
* Active autoimmune diseases requiring systemic treatment (such as the use of disease relieving drugs, glucocorticoids or immunosuppressants) occurred within 2 years before the first administration. Alternative therapy (such as thyroxine, insulin or physiological glucocorticoid for adrenal or pituitary insufficiency) is not considered as systemic therapy;
* The study was receiving systemic glucocorticoid treatment (excluding local glucocorticoids by nasal spray, inhalation or other means) or any other form of immunosuppressive therapy within 7 days before the first administration;
* Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* People known to be allergic to the drugs used in this study;
* People with multiple factors affecting capecitabine (such as inability to swallow and intestinal obstruction);
* Before starting treatment, the patient has not fully recovered from the toxicity and/or complications caused by any intervention (i.e. ≤ Level 1 or reaching the baseline, excluding fatigue or hair loss);
* Known history of human immunodeficiency virus (HIV) infection (i.e. HIV /2 antibody positive);
* Untreated active hepatitis B ；
* Active HCV infected subjects；
* Live vaccine shall be inoculated within 30 days before the first administration (the first cycle, the first day);
* Pregnant or lactating women;
* Abnormal medical history or disease evidence, treatment or laboratory test value that may interfere with the test results, prevent the subject from participating in the study in the whole process, or other conditions that the researcher believes are not suitable for inclusion. The researcher believes that there are other potential risks that are not suitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 7 days after surgery
  Pathological remission rate according to Becker standard

SECONDARY OUTCOMES:
MPR | 7 days after surgery
  major pathologic response according to Becker standard
DFS | Long term follow-up will continue until the death of the subject or the end of the study, at least three years
  disease-free survival
R0 resection rate | postoperative 6 hours
  Proportion of R0 level surgery performed
OS | Long term follow-up will continue until the death of the subject or the end of the study, at least three years
  overall survival
ORR | 7 days after surgery
  Objective remission rate
Adverse reactions and perioperative complications (Security) | Long term follow-up will continue until the death of the subject or the end of the study, at least three years
  Adverse reactions and perioperative complications caused by drug therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Wang Nan, Xi’an, Shanxi, China